CLINICAL TRIAL: NCT05933291
Title: Single-cell Landscape of BALF in Patients With Severe ARDS and CARDS: an Analysis of the Effectiveness of Steroid Therapy and a Comparison Between COVID-19 ARDS and ARDS From Other Etiologies
Brief Title: Single-cell Landscape of BALF in Patients With Severe ARDS and CARDS
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Covid20230601
Record Dates: First submitted 2023-06-02; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: ARDS: Acute Respiratory Distress Syndrome; Covid19
MeSH Terms: conditions — Acute Lung Injury; COVID-19 | interventions — Steroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — BALF
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- COVID-19 with steroid: COVID-19 ARDS patients with steroid treatment
  Interventions: Drug: steroid
- COVID-19 without steroid: COVID-19 ARDS patients without steroid treatment
- non-COVID-19 with steroid: non-COVID-19 ARDS patients with steroid treatment
  Interventions: Drug: steroid
- non-COVID-19 without steroid: non-COVID-19 ARDS patients without steroid treatment

INTERVENTIONS:
Drug: steroid — Moderate- or high-dose steroids
  Groups: COVID-19 with steroid; non-COVID-19 with steroid

SUMMARY:
The goal of this observational study is to learn about the effect of steroid therapy in patients with COVID-19 ARDS. The main questions it aims to answer are:

* Differences between patients with COVID-19 ARDS before and after steroid treatment in BALF single cell landscape, as well as patients with different prognosis.
* Differences between COVID-19 and non COVID-19 ARDS patients in BALF single cell landscape.

Participants will Choose whether to use or not to utilize steroid treatment based on conditions.

DETAILED DESCRIPTION:
Collect BALF from COVID-19 and non-COVID-19 ARDS patients both before and during remission, then perform single-cell sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Severe ARDS patients

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 4 COVID-19 ARDS patients, 4 non-COVID-19 ARDS patients
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-09-24 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
single-cell analysis in BALF before treatment | before treatment in ICU
  collect BALF before and during treatment and perform single-cell sequencing
single-cell analysis in BALF after treatment | After treatment in ICU for 1-4 weeks
  collect BALF before and during treatment and perform single-cell sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Yun Long, MD, Study Director — Peking union medical college hospital, ICU department
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China